CLINICAL TRIAL: NCT02210455
Title: Strongest Families FASD: Parent Training for Challenging Behaviour in Children With Fetal Alcohol Spectrum Disorder (FASD)
Brief Title: Parenting Training for Children With FASD
Acronym: SF-FASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Collaborators: NeuroDevNet (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Queen's University (Other); Public Health Agency of Canada (PHAC) (Other Government)
Responsible Party: Principal Investigator, Patrick J. McGrath, Integrated Vice President Research and Innovation, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1017014
Record Dates: First submitted 2014-07-30; First posted 2014-08-06 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Fetal Alcohol Spectrum Disorder
Keywords: FASD; pFAS; ARND; Fetal Alcohol Syndrome; Partial Fetal Alcohol Syndrome; Alcohol Related Neurodevelopmental Disorder; Static Encephalopathy (Alcohol Exposed); Neurobehavioural Disorder (Alcohol Exposed)
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Strongest Families FASD intervention (Experimental): It is a web-based parent training program with a coach. The program is comprised of 11 sessions, each focusing on a different parenting strategy, delivered using easy to read text, instructional videos and audio clips. One Booster Session is conducted 1 month after completion of Session 11.
  Interventions: Behavioral: Strongest Families FASD intervention; Other: Psychoeducation
- Psychoeducation (Active Comparator): It is a static webpage on IRIS providing FASD information and resources, including recommended book titles, websites and organizations that may be helpful.
  Interventions: Other: Psychoeducation

INTERVENTIONS:
Behavioral: Strongest Families FASD intervention
  Arms: The Strongest Families FASD intervention
Other: Psychoeducation

SUMMARY:
Prenatal alcohol exposure can lead to a myriad of adverse developmental outcomes in children, and is the leading cause of mental disability in Canada. The term fetal alcohol spectrum disorders (FASD) was established to encompass the full spectrum of teratogenic effects induced by alcohol. FAS is believed to occur in approximately 1 to 3 per 1000 live births in North America, and it is estimated that FASD may occur as frequently as 1 in 100 live births, making this a public health problem of epidemic proportion. Even though considerable efforts have been aimed at identifying children with FASD, the need for access to services and supports for Canadian families affected by FASD remains unfulfilled. Additionally, there is little empirical data available to influence policy change in how these services and supports are delivered.

A key recommendation contained in the Public Health Agency of Canada's (PHAC) Fetal Alcohol Spectrum Disorder (FASD): A Framework for Action document was the need to determine the types of supports children with FASD and their families require and to develop appropriate mechanisms to provide these services at the community, provincial/territorial and federal levels. This identified need forms the basis of the current proposal.

Although a variety of psychosocial interventions have been developed to treat neurobehavioural disorders, relatively little research has been conducted that is specifically aimed at improving the behavioral challenges identified in children with FASD. Thus, we hypothesize that (i) a FASD-specific parent/guardian training intervention can be developed using input from major stakeholders to meet the current limitations in access for families seeking services and supports; and (ii) this intervention and its evaluation will provide evidence for feasibility and efficacy to support changes in policy by key decision-makers and provide the basis for developing promising practices in the area of interventions for families affected by FASD. This grant will link academic teams with parents/guardians and decision makers to develop and evaluate a training program for the parents/guardians of children with FASD.

Participants will be recruited from across Canada. The specific objectives of the proposed research program, which will be addressed in three inter-related studies, are to:

1. Develop an Internet-based intervention program for parents/guardians of children with FASD between the ages of 4-12 years, that is based on information collected from interviews completed by major stakeholders (e.g., parents/guardians, clinicians, decision-makers, community-based organizations);
2. Evaluate the feasibility (usability) of the intervention; and
3. Obtain data on outcomes from the randomized controlled trial This research will adopt an integrated knowledge translation and exchange approach where knowledge production, dissemination, uptake and usage will occur seamlessly throughout the project and researchers and knowledge users are engaged in the project right from its inception.

The intervention will be based on the Strongest Families program that is designed to help families learn to deal with common childhood problems in the comfort and privacy of their home, and provide treatment and care via telephone contact with trained coaches, written manuals, videotapes, and audiotapes. This program has been successful in children neurodevelopmental disorders; and will be adapted for use in the FASD population, as children with FASD, share many of the same behavioral characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Have a child between 4-12 years of age with a diagnosis which falls under the umbrella term "Fetal Alcohol Spectrum Disorder" as reported by parents/caregivers.
* The child has been experiencing behavioural problems (as defined by the caregiver) for at least 6 months prior to study screening.
* Have been the primary caregiver for a minimum of 6 months prior to entry into the study.
* Have a reasonable expectation of being be the primary caregiver for at least 6 months after study enrolment.
* Read, write, and understand English.
* Have access to a telephone.
* Have access to a computer connected to the Internet.
* Live in Canada.
* CBCL Externalizing t-Score must be ≥64 (clinical range)
* The child meets criteria for behaviour suggestive of FASD
* No suicide attempts within the previous 6 months
* No current risk of suicide attempts

Exclusion Criteria:

* Child is NOT able to speak in full sentences or understand everyday language and instructions.
* Parent/caregiver has previously taken part in a Strongest Families Parenting Program.
* Parent/caregiver OR child has been diagnosed with Psychosis.
* Child does not have a diagnosis of schizophrenia, bipolar disorder or major depression.
* Child does not put others as risk of serious harm (i.e., requiring medical attention).
* Parent/caregiver has not completed any of the following parenting programs in the last 6 months: Triple P, COPE, Incredible Years.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
A change on the Child Behavior Checklist from baseline to 11 months | At baseline, and 5 months and 11 months after randomization
  It is a standardized questionnaire that assesses adaptive functioning and problems. We will use two versions of the CBCL (CBCL/1 ½ -5 and CBCL/6-18) to accommodate the age range of the sample

SECONDARY OUTCOMES:
A change on the Depression Anxiety & Stress Scale Short Form (DASS-21) from baseline to 11 months | At baseline, and 5 months and 11 months after randomization
  It will be used to evaluate parental distress
Client Satisfaction Questionnaire (CSQ-8) | Participants will be asked to complete this measure at the end of the intervention, which will probably last on average 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McGrath, PhD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be shared.

REFERENCES:
- [Derived] Turner K, Reynolds JN, McGrath P, Lingley-Pottie P, Huguet A, Hewitt A, Green C, Wozney L, Mushquash C, Muhajarine N, Sourander A, Caughey H, Roane J. Guided Internet-Based Parent Training for Challenging Behavior in Children With Fetal Alcohol Spectrum Disorder (Strongest Families FASD): Study Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2015 Oct 13;4(4):e112. doi: 10.2196/resprot.4723. PMID 26462968